CLINICAL TRIAL: NCT02206178
Title: ACETAMINOPHEN ANTINOCICEPTIVE EFFECT WHEN ASSOCIATED WITH N-ACETYLCYSTENEINE
Brief Title: Acetaminophen's Antinociceptive Effect When Associated With N-Acetylcysteneine
Acronym: PANACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0202; 2013-000668-27
Record Dates: First submitted 2014-07-29; First posted 2014-08-01 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- acetaminophen (Experimental): The purpose of this study is to assess the effectiveness of acetaminophen in association with N-acetylcysteine.
  The objective of this study is to evaluate if the association in healthy volunteers of acetaminophen and N-acétylcystéine
  1. - decrease the antinociceptive effect of acetaminophen in comparison to a group control
  2. - and if this antinociceptive effect may depend of the genetic polymorphism of GSH enzyme
  Interventions: Drug: N-acetylcysteine combination with acetaminophen
- placebo (Placebo Comparator): 1. - decrease the antinociceptive effect of acetaminophen in comparison to a group control
  2. - and if this antinociceptive effect may depend of the genetic polymorphism of GSH enzyme
  Interventions: Drug: N-acetylcysteine combination with acetaminophen; Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine combination with acetaminophen
Drug: Placebo
  Arms: placebo

SUMMARY:
Acetaminophen is one of the most widely used analgesic in the world, recommended for the symptomatic treatment of fever and pain.

The purpose of this study is to assess the effectiveness of acetaminophen in association with N-acetylcysteine.

The objective of this study is to evaluate if the association in healthy volunteers of acetaminophen and N-acétylcystéine

1. - decrease the antinociceptive effect of acetaminophen in comparison to a group control
2. - and if this antinociceptive effect may depend of the genetic polymorphism of GSH enzyme.

DETAILED DESCRIPTION:
Period 1 : To Day -4 to Day 0

Day -4 at 8:00 am at Clinical Pharmacology Center

* Inclusion Visit, signature of Informed consent form, clinical exam.
* Training test
* Blood sample (GSH, pharmacogenetic, Biochemistry assay)
* Randomization and attribution of treatment for the fisrt study period at home: (day -4, -3, -2, -1) 4 days of oral acetaminophen and [N-acetylcysteine or placebo] according to the randomization plan.

At day -3, -2 and -1 a salivary sample will be done to control the treatment compliance.

Day 0 at Clinical Pharmacology Center Clinical examination Measurement of the basal pain thresholds and pain evaluation (Visual Analog Scales) Blood and urinary sample (acetaminophen and GSH assay)

T0 : Administration of product: acetaminophen and [N-acetylcysteine or placebo]

T0+1H: Thermal stimulation according to the established paradigm (threshold temperature +3°C ) and pain evaluation (Visual Analog Scales)

T0+2H: Thermal stimulation according to the established paradigm (threshold temperature +3°C ) and pain evaluation (Visual Analog Scales) and Blood sample (acetaminophen assay)

T0+3H: Thermal stimulation according to the established paradigm (threshold temperature +3°C ) and pain evaluation (Visual Analog Scales)

T0+4H: Thermal stimulation according to the established paradigm (threshold temperature +3°C ) and pain evaluation (Visual Analog Scales) and Blood and urinary sample (acetaminophen, GSH, biochemistry assay)

- Lunch before departure

2 weeks of wash-out

Period 2 : To Day 17 to Day 21

Same of period 1. Subject who receives N-acétylcystéine in period 1 will receive placebo in second period and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between 18 and 45 years old
* Without treatment during the 7 days before inclusion specially no use of antalgic and anti-inflammatory
* Cooperation and understanding enough to conform to the study obligations -Having given free, informed written consent
* Affiliated at system of French social security
* Inscription or acceptation of inscription in the national register of volunteers involved in trials.

Exclusion Criteria:

* Patient with one or many contraindication for the administration of the trial's products,
* Patient that have taken N-acetylcysteine as bronchial thinner during the last 3 days,
* Patient with medical or surgical history judged by the investigator or his representative as being not compatible with the clinical trial
* Patient with disease progression during inclusion,
* Patient with excessive consumption of alcohol, tobacco (+ than 10 cigarette/day), coffee, tea or drinks with caffeine (equivalent to more than 4 cup a day) or any addiction to drugs,
* Patient with a heat pain mean threshold during training higher or equal to 46.5°C,
* Patient who participated in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial,
* Patient with cooperation and understanding that do not allow him to follow the trial,
* Patients with minor or under guardianship,
* No affiliation at system of French social security

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity using Visual Analog Scales (VAS) succeeding thermic stimulations at the threshold temperature +3°C before (T0-1h) and after acetaminophen's administration | At day 0
  Pain intensity using Visual Analog Scales (VAS) succeeding thermic stimulations at the threshold temperature +3°C before (T0-1h) and after acetaminophen's administration (T0+1h, T0+2h, T0+3h, T0+4h).

SECONDARY OUTCOMES:
Blood glutathione GSH concentration | At day 0
  Blood glutathione GSH concentration at J0 T0-1h and J0 T0+4h
Blood of acetaminophen concentration and its metabolites | at day 0
  Blood of acetaminophen concentration and its metabolites at J0 T0-1h, T0+2h, and T0+4h.
Urinary assay of the rate of acetaminophen and its metabolites | at day 0
  Urinary assay of the rate of acetaminophen and its metabolites at J0 T0-1h, and T0+4h.
Pharmacogenetic dosage of enzymes involved in glutathione metabolism | at day 4

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France